CLINICAL TRIAL: NCT07187037
Title: Comparison of the Effects of the Interaction of Methylprednisolone and Dexamethasone With Sugammadex on Rocuronium Reversal Time, Postoperative Pain, and Nausea in Adult Patients
Brief Title: Methylprednisolone vs Dexamethasone: Effects on Sugammadex Reversal, Pain, and Nausea in Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, MUSTAFA BÜYÜKCAVLAK, Specialist in Anesthesiology and Intensive Care, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AEŞH-EK-2025- 100
Record Dates: First submitted 2025-09-11; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Neuromuscular Block, Residual; Pain; Postoperative Nausea
Keywords: sugammadex; dexamethasone; methylprednisolone; postoperative nausea; postoperative pain
MeSH Terms: conditions — Delayed Emergence from Anesthesia; Pain; Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Methylprednisolone; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylprednisolone Group (Active Comparator): Patients will receive intravenous methylprednisolone 1 mg/kg diluted in 5 mL saline, administered at anesthesia induction.
  Neuromuscular blockade will be achieved with rocuronium.
  Reversal will be performed with sugammadex 2 mg/kg at reappearance of the second twitch in train of four monitoring.
  Interventions: Drug: Methylprednisolone (MP)
- Dexamethasone Group (Active Comparator): Patients will receive intravenous dexamethasone 0.2 mg/kg diluted in 5 mL saline, administered at anesthesia induction.
  Neuromuscular blockade will be achieved with rocuronium.
  Reversal will be performed with sugammadex 2 mg/kg at reappearance of second twitch in train of four monitoring
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Methylprednisolone (MP) — Methylprednisolone 1 mg/kg IV (diluted to 5 mL with saline) will be administered at induction of anesthesia. Neuromuscular blockade will be achieved with rocuronium. Reversal will be performed with sugammadex 2 mg/kg IV at the reappearance of the second twitch in train of four monitoring.
  Arms: Methylprednisolone Group
Drug: Dexamethasone — Dexamethasone 0.2 mg/kg IV (diluted to 5 mL with saline) will be administered at induction of anesthesia. Neuromuscular blockade will be achieved with rocuronium. Reversal will be performed with sugammadex 2 mg/kg IV at the reappearance of second twitch in train of four monitoring.
  Arms: Dexamethasone Group

SUMMARY:
This randomized controlled trial aims to compare the effects of intravenous methylprednisolone and dexamethasone on the reversal time of rocuronium by sugammadex in adult patients undergoing elective septoplasty or rhinoplasty. The primary outcome is the time from sugammadex administration to recovery of a train-of-four (TOF) ratio of 0.9. Secondary outcomes include extubation time, postoperative nausea and vomiting (PONV), pain scores, complications in the post-anesthesia care unit (PACU), and intraoperative hemodynamic parameters. The study will provide new evidence on whether perioperative corticosteroid choice modifies the efficacy of sugammadex and influences postoperative recovery.

DETAILED DESCRIPTION:
Neuromuscular blockade with rocuronium is routinely reversed with sugammadex. Corticosteroids such as methylprednisolone and dexamethasone are frequently used perioperatively for their anti-inflammatory and antiemetic effects. However, possible pharmacological interactions between corticosteroids and sugammadex remain unclear and may affect reversal time.

This prospective, randomized, parallel-group clinical trial will enroll adult ASA I-II patients scheduled for elective septoplasty or rhinoplasty. Patients will be randomized to receive either methylprednisolone (1 mg/kg IV) or dexamethasone (0.2 mg/kg IV) at induction of anesthesia. Rocuronium will be administered for neuromuscular blockade, and sugammadex (2 mg/kg IV) will be given at the reappearance of the second twitch in TOF monitoring. Neuromuscular recovery will be continuously assessed with acceleromyography at the adductor pollicis muscle.

The primary outcome is the time interval from sugammadex injection to a TOF ratio of 0.9.

Secondary outcomes include extubation time, total rocuronium consumption, incidence and severity of PONV (assessed by VAS-B at 0, 30, 60, and 120 minutes in PACU), postoperative pain (VAS-A at the same time points), PACU complications (desaturation, stridor, severe cough), and intraoperative hemodynamic variables.

All anesthetic procedures will be standardized, and outcome assessors and statisticians will be blinded to group allocation. The results of this trial may guide perioperative steroid selection in patients receiving sugammadex reversal and help optimize postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-65 years
* American Society of Anesthesiologists (ASA) physical status I-II
* Scheduled for elective septoplasty or rhinoplasty under general anesthesia
* Written informed consent obtained

Exclusion Criteria:

* ASA physical status ≥ III
* Emergency surgery
* Known allergy or contraindication to rocuronium, sugammadex, or corticosteroids
* Chronic or recent (within 3 months) systemic corticosteroid therapy
* Concomitant use of drugs that may interact with sugammadex (e.g., toremifene, flucloxacillin, fusidic acid)
* Neuromuscular disorders (e.g., myasthenia gravis, muscular dystrophy)

  * Significant hepatic, renal, respiratory, or cardiac dysfunction
* Anticipated difficult airway or history of difficult intubation
* Nasopharyngeal or oropharyngeal anomalies interfering with airway management
* Developmental or cognitive impairment interfering with informed consent or cooperation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Reversal Time | Perioperative period (Immediately after sugammadex administration until achievement of a normalised train-of-four ratio ≥0.9, measured in seconds)
  The interval in seconds between intravenous administration of sugammadex (2 mg/kg) and achievement of a normalised train-of-four ratio ≥0.9 measured at the adductor pollicis muscle using acceleromyography.

SECONDARY OUTCOMES:
Extubation time | Perioperative period (from sugammadex administration until tracheal extubation, in minutes)
  Time in minutes from sugammadex injection to tracheal extubation in perioperative period.
Postoperative pain scores | At 2 hours postoperatively
  Pain intensity assessed with Visual Analogue Scale for Pain (VAS-A; 0-10 scale).
Postoperative nausea and vomiting (PONV) incidence and severity | At 2 hours postoperatively
  Presence and severity of nausea and vomiting, assessed using Visual Analogue Scale for Nausea and Vomiting (VAS-B; 0-10 scale).

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Karatay, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zwiers A, van den Heuvel M, Smeets J, Rutherford S. Assessment of the potential for displacement interactions with sugammadex: a pharmacokinetic-pharmacodynamic modelling approach. Clin Drug Investig. 2011;31(2):101-11. doi: 10.2165/11584730-000000000-00000. PMID 21067251
- [Background] Fortier LP, McKeen D, Turner K, de Medicis E, Warriner B, Jones PM, Chaput A, Pouliot JF, Galarneau A. The RECITE Study: A Canadian Prospective, Multicenter Study of the Incidence and Severity of Residual Neuromuscular Blockade. Anesth Analg. 2015 Aug;121(2):366-72. doi: 10.1213/ANE.0000000000000757. PMID 25902322